CLINICAL TRIAL: NCT05646095
Title: B-SAFE: A Trauma-Informed Early Intervention Targeting Sleep and Adjustment Among Children in Foster Care
Brief Title: A Trauma-Informed Sleep Intervention for Children in Foster Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Candice A Alfano (Other)
Responsible Party: Sponsor-Investigator, Candice A Alfano, Professor, University of Houston
Organization: University of Houston (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 000181698
Record Dates: First submitted 2022-02-21; First posted 2022-12-12 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Sleep Disturbance; Child Development; Mental Disorder, Child
MeSH Terms: conditions — Parasomnias; Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: multi-phase hybrid effectiveness-implementation trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolstering Sleep and Adjustment in Foster Environments (B-SAFE) (Experimental): Brief, behavioral sleep intervention for children and caregivers
  Interventions: Behavioral: Bolstering Sleep and Adjustment in Foster Environments (B-SAFE)
- Delayed Intervention (Active Comparator): Waitlist families will be monitored for 1 month before receiving the B-SAFE intervention
  Interventions: Behavioral: Bolstering Sleep and Adjustment in Foster Environments (B-SAFE)

INTERVENTIONS:
Behavioral: Bolstering Sleep and Adjustment in Foster Environments (B-SAFE) — We will adapt CBT for insomnia for children in foster care using a trauma-informed approach that considers the child's individual history, unique family environment, and child welfare policies regarding safe sleep practices.

SUMMARY:
Sleep disturbances are pervasive and impairing among children who spend time in foster care but not a single prevention or intervention program for this fragile group targets sleep health. Poor sleep undermines effective self-regulation and stable biological rhythms, amplifying the negative impacts of early adversity/trauma on immediate and long-term functioning. Consistent with evidence that optimizing sleep is critical for trauma recovery, the investigators will adapt cognitive-behavioral treatment for pediatric insomnia for children placed in or adopted from foster care to evaluate child outcomes and target mechanism engagement and explore implementation barriers and supports.

DETAILED DESCRIPTION:
Children in foster care (FC) evidence poorer developmental, physical and mental health outcomes than even the poorest children in the U.S. and unmet need in this fragile group is extraordinarily high. Of the small number of early intervention programs demonstrated as effective for this population, most are directed at infants and young children. However, more than half of the children entering FC each year are older than 5 years, a time when capacity for and expectations of self-regulation are greater, but history of maltreatment/trauma is often more extensive.

Sleep disturbance is one of the most well-recognized consequences and enduring sequela of early adversity/trauma that creates a feedback loop through which arousal/anxiety is amplified, self-regulation is undermined, and biological rhythms are altered. Mounting evidence reveals behavioral sleep problems to be prevalent among a majority of children in FC and closely associated with elevated mental health problems. Early intervention programs targeting sleep might therefore prevent a cascade of negative outcomes and serve to reduce placement disruption risk.

The research team, with unique expertise in pediatric sleep, childhood maltreatment, attachment, and the delivery of foster care interventions, will use a trauma-informed framework to adapt cognitive-behavioral therapy for pediatric insomnia for school-aged children in and adopted from FC. A 3-year, multi-phase hybrid effectiveness-implementation trial will: a) determine whether the intervention, Bolstering Sleep and Adjustment in Foster Environments (B-SAFE) has measurable effects on the sleep, emotional and behavioral health of children (6 to 10 years) in or adopted from foster care; and b) engage stakeholders early in the implementation process to ensure alignment of the B-SAFE program with child welfare resources and family needs. B-SAFE's target mechanisms are informed by research showing reductions in children's nighttime anxiety/arousal and increased parental support around bedtime/sleep routines to correspond with better child sleep, emotional and behavioral health. Phase 1 will include input and feedback from FC agency partners in the local community, expert consultants, and pilot families in order to finalize the intervention manual, materials, and procedures. In Phase 2, the investigators will conduct a randomized, controlled trial among N=60 new families; 30 will receive the B-SAFE right away and 30 will serve as waitlist (WL) controls. Post treatment and follow up assessments of child sleep health, emotional/behavioral regulation, and biological rhythms will be examined via objective and subjective measures. In the last year of the project, the investigators will conduct quantitative surveys and qualitative interviews with key stakeholders to explore potential barriers to and available supports/resources for a larger implementation trial.

ELIGIBILITY:
Inclusion Criteria:

1. All non-relative foster, kinship and adoptive foster families with a child between the ages 6 and 10 years who have been in the home for one month.
2. A caregiver or child-reported behavioral sleep problem at least twice a week.

Exclusion Criteria:

1. Children who are considered 'medically fragile' or with serious medical issues/conditions requiring routine care, supervision/monitoring and/or regular use of equipment (e.g., paralysis, tracheostomy, blindness, cerebral palsy). We will not exclude children with non-serious medical conditions that are well-managed (e.g., asthma, diabetes, HIV).
2. Children with significant developmental delays or intellectual disability who would have difficulty comprehending and/or engaging in treatment. Consistent with practices in community settings, the study team will consider the reliability of child responses during the initial assessment to identify children who meet this criterion (rather than standardized test scores).
3. Children with a confirmed or suspected medical sleep disorder requiring medical treatment (e.g., obstructive sleep apnea, narcolepsy). We will immediately refer these children for services as necessary.
4. Foster parent and/or child who is a non-fluent English speaker.
5. Current foster parent or child suicidality or self-harm behaviors (i.e., suicidal ideation, intent, and/or plan, cutting, burning, etc).

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Child average total sleep time (TST) | one week and 3-months follow up
  Changes in TST will be assessed using subjective sleep logs and wrist actigraphy across one week
Child average wake minutes after sleep onset (WASO) | one week and 3-months follow up
  Changes in WASO will be assessed using subjective sleep logs and wrist actigraphy across one week
Child average sleep onset latency (SOL) | one week and 3-months follow up
  Changes in SOL will be assessed using subjective sleep logs and wrist actigraphy across one week
Change in Emotional and behavioral regulation | one week and 3-months follow up
  Reports on the NIH Toolbox Emotion Control measure will be used to assess changes in emotional and behavioral regulation. Difference in subjective reports on the NIH Toolbox Fixed Form v2.0 - Emotion Control v2.0 Measure will be compared at baseline (week 0) and post treatment (3 months later). The raw score is calculated by summing up the 10 items in the measure. Raw scores are converted to Toolbox Age-Adjusted, Fully Adjusted and Unadjusted Scale Scores for PROs - Mean of 50, SD of 10. Higher scores are an indicative of greater emotional regulation and lower scores are indicative of lower levels of emotional regulation.
Cortisol awakening response (mcg/dL) | one week and 3-months follow up
  Changes in biological rhythms will be assessed via morning and evening salivary cortisol across two non-consecutive days during the same week
Objective sleep timing (mid sleep point) | one week and 3-months follow up
  Changes average mid sleep point across across one week based on actigraphy

SECONDARY OUTCOMES:
Pre-Sleep Arousal Scale for Children (PSAS-C) | one week and 3-months follow up
  Difference in subjective reports of children on Pre-Sleep Arousal Scale for Children (PSAS-C) measure will be compared at baseline (week 0) and post treatment (3 months later). The raw score is calculated by summing up the 16 items in the measure with scores ranging from 16 to 80. Higher scores indicate higher states of arousal before sleep.
Children's Sleep Habits Questionnaire (CSHQ) | one week and 3-months follow up
  Difference in subjective reports of parents on Children's Sleep Habits Questionnaire (CSHQ) measure will be compared at baseline (week 0) and post treatment (3 months later). The measure produces 8 subscales: bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night awakening, parasomnias sleep disordered breathing, and daytime sleepiness. The subscales are scored by summing up the score of all items' in a subscale. The total sleep disturbance score is the sum of all the subscales, with higher scores indicating more sleep disturbances.
Bedtime Routines Questionnaire (BRQ) | one week and 3-months follow up
  Difference in subjective reports of parents on The Bedtime Routines Questionnaire will be compared at baseline (week 0) and post treatment (3 months later). The Bedtimes Routines Questionnaire produces 4 subscales: total reactivity, total consistency, adaptive and maladaptive activity. Each subscale is calculated by summing the items compromising the subscales. Greater scores suggest greater reactivity to changes in routine (range 5 to 25), greater routine consistency (range 10 to 50) and more frequent adaptive (range 10 to 50) and maladaptive activities (range 6 - 30).

OTHER OUTCOMES:
Rates of retention | 3-months follow up
  Treatment Feasibility will be assessed based on rates of retention/attrition during the study. Treatment feasibility will be assessed based on the retention during the study. The retention rate is defined as the percentage of participants who complete the study.
Rates of attrition | 3-months follow up
  Treatment feasibility will be assessed based the attrition rate during the study. The attrition rate is defined as the percentage of participants who drop out of the study.
Homework Compliance | one week
  Treatment feasibility will be assessed based on homework compliance during treatment. Homework compliance is defined as the percentage of completed homework assignments compared to the total number of assigned homework.
Client Satisfaction Questionnaire (CSQ) | one week
  Treatment acceptability will be accessed based on the ratings using the Client Satisfaction Questionnaire (CSQ). The CSQ is an 8-item measure scored on a 4 point Likert scale. The sum of the items produces a total score, ranging from 8 to 32. Higher scores indicate greater client satisfaction.
Parenting Stress Index -Short Form (PSI) | one week and 3-months follow up
  Changes in parenting Stress will be assessed using the PSI. Difference in subjective reports on Parenting Stress Index -Short Form will be compared at baseline (week 0) and post treatment (3 months later). The measure produces 3 subscales: parental distress, parent- child dysfunctional interaction and difficult child. The total score is the sum of the three subscales. Higher scores indicate higher levels of stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep and Anxiety Center of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes